CLINICAL TRIAL: NCT05012527
Title: Retrospective Review of Gastrointestinal System Endoscopy Procedures
Acronym: RRGIE
Status: Completed | Type: Observational
Sponsor: Istanbul Sultanbeyli State Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammer Ergenç, MD, General Surgeon, Istanbul Sultanbeyli State Hospital
Other Study IDs: 2021s01
Record Dates: First submitted 2021-07-15; First posted 2021-08-19 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Endoscopy; Colonoscopy; Gastroscopy; Colonic Polyps; Endoscopy, Digestive System; Gastrointestinal Neoplasms; Biopsy
MeSH Terms: conditions — Colonic Polyps; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is retrospectively evaluating all features of endoscopic and pathological diagnoses of cases who underwent upper and lower gastrointestinal endoscopy.

DETAILED DESCRIPTION:
Gastrointestinal system endoscopy has an important place in the diagnosis and treatment of many diseases related to this system and provides an alternative to current surgical methods with its ever-expanding field of application. Upper and lower gastrointestinal endoscopy procedures are performed with many indications, such as new complaints in the gastrointestinal tract at the age of 50 and over, family history of gastrointestinal malignancy. In addition, the importance of endoscopy is gradually increasing as tissue and cell samples can be taken for histopathological studies and endoscopic treatment of some diseases.

The aim of the study is to review patients' indications, distribution by age and gender, frequency of lesions diagnosed on endoscopy, prevalence, size, histology and location of polyps detected and excised, results of endoscopic and pathological diagnoses.

The study population consists of the patients who were examined at the Istanbul Sultanbeyli State Hospital Endoscopy Unit between 01.01.2016 and 01.01.2021.

The patients' data will be scanned retrospectively by accessing their files from the computer database.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old)
* Patients who have undergone the procedure in our endoscopy unit

Exclusion Criteria:

* Under 18 years old
* Patients whose information cannot be accessed in the system records.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of the patients who were examined at the Istanbul Sultanbeyli State Hospital Endoscopy Unit between 01.01.2016 and 01.01.2021.
Sampling Method: Non-Probability Sample
Enrollment: 15448 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Age | During 3 months (retrospective endoscopy data review)
  Age distribution of patients in endoscopic procedures and histopathological examinations
Gender | During 3 months (retrospective endoscopy data review)
  Sex distribution of patients in endoscopic procedures and histopathological examinations
Type of endoscopy | During 3 months (retrospective endoscopy data review)
  Number of each endoscopy, Type (esophagogastroduodenoscopy, colonoscopy, rectosigmoidoscopy)
Indications | During 3 months (retrospective endoscopy data review)
  Number of endoscopic indications, Type (Abnormal imaging, GI bleeding, Anemia, Screening and surveillance, Diarrhea, Constipation, Abdominal pain, Weight loss, Dyspepsia, Heartburn, Dysphagia, Odynophagia, Upper belly pain or chest pain that is not heart-related, Intractable vomiting, Bleeding in the upper, Persistent gastroesophageal reflux symptoms, Occult gastrointestinal bleeding, Other)
Procedure-related complications rates | During 3 months (retrospective endoscopy data review)
  The patients with complications / the total patients
  Number of adverse events; early or late (within 1 month), related to the endoscopic procedure, Type (cardiopulmonary complication, gastrointestinal bleeding, perforation, mortality)
Prevalence of benign/malign gastrointestinal disease in the endoscopy | During 3 months (retrospective endoscopy data review)
  The patients with benign gastrointestinal disease / the total patients
  The patients with malign gastrointestinal disease / the total patients
Polyp/tumor detection rate of screening endoscopy | During 3 months (retrospective endoscopy data review)
  The patients with polyp / the total number of screening endoscopy patients
  The patients with tumor / the total number of screening endoscopy patients
Polyp/tumor detection rate of symptomatic patients' endoscopy | During 3 months (retrospective endoscopy data review)
  The patients with polyp / the total number of symptomatic patients endoscopy
  The patients with tumor / the total number of symptomatic patients endoscopy
Polyps localization and frequency | During 3 months (retrospective endoscopy data review)
  The patients with polyp / the total patients
  Number of polyp localizations, Type (Rectum, Sigmoid colon, Descending colon, Splenic flexure, Transverse colon, Hepatic flexure, Ascending colon, Caecum, Multiple localization)
Non-neoplastic biopsy results | During 3 months (retrospective endoscopy data review)
  The patients with non-neoplastic biopsy results / the total patients
Prevalence of gastric/bowel diseases in histopathology | During 3 months (retrospective endoscopy data review)
  The patients with gastric disease / the total patients
  The patients with bowel disease / the total patients
Prevalence of advanced neoplasia | During 3 months (retrospective endoscopy data review)
  The patients with advanced neoplasia / the total patients
Prevalence of gastric/colorectal cancer | During 3 months (retrospective endoscopy data review)
  The patients with gastric cancer / the total patients
  The patients with colorectal cancer / the total patients
Completeness rate of the procedures | During 3 months (retrospective endoscopy data review)
  The number of completed procedures / total number of procedures

CONTACTS AND LOCATIONS:
Overall Officials: Muhammer Ergenç, MD, Principal Investigator — Istanbul Sultanbeyli State Hospital
Locations (1):
- Istanbul Sultanbeyli State Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided